CLINICAL TRIAL: NCT00181129
Title: Mitigating Cancer Treatment-Related Fatigue by Exercise
Brief Title: Fatigue and Cancer Treatment(FACT)- an Exercise Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NINR:RO1NRO4991
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Cancer; Fatigue
Keywords: Fatigue; Cancer treatment
MeSH Terms: conditions — Neoplasms; Fatigue

INTERVENTIONS:
Behavioral: home based self paced walking program

SUMMARY:
The purpose of this randomized controlled trial is to determine the effects of a nurse-directed, home-based walking exercise program to mitigate fatigue and maintain physical functioning during adjuvant therapy for cancer. The sample will be randomized into exercise (EX) or usual care (UC) groups. The independent study variable is participation in a walking exercise program. Outcomes include: fatigue, sleep disturbance, emotional distress, physical functioning and quality of life. The effects of the walking exercise program will be evaluated using self-report questionnaires administered pre- and post-treatment, patient diaries, and symptoms assessments at defined intervals during adjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of cancer (Stage 1,2,or 3),

21 years of age or older,

Free of cognitive or physical deficits that would preclude entry into study,

not currently exercising 120 min/wk or more

Exclusion Criteria:

Concurrent major health problems or disabilities that would limit participation in an exercise program.

Stage 4 cancer (metastisis)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2002-09 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria L Mock, DNSc, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins University School of Nursing, Baltimore, Maryland, United States